CLINICAL TRIAL: NCT01200836
Title: Effects of Rosuvastatin on the Immune System in Healthy Volunteers With Normal Cholesterol
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100165; 10-H-0165
Record Dates: First submitted 2010-09-10; First posted 2010-09-14 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10-04

CONDITIONS: Healthy Volunteers; Statins; Immune Modulation
Keywords: Statins; Immune Modulation; Healthy Volunteer

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- The drug rosuvastatin (also called Crestor) is used to lower cholesterol levels in people with elevated cholesterol levels. Recent studies have suggested that rosuvastatin may affect the immune system and reduce inflammation, but the reason for this effect is unclear. Researchers are interested in testing the effect of rosuvastatin on the immune systems of healthy volunteers with good cholesterol levels.

Objectives:

- To evaluate the effect of rosuvastatin on the immune systems of healthy volunteers.

Eligibility:

- Healthy individuals at least 18 years of age who have an acceptable blood level of LDL cholesterol (below 160).

Design:

* Participants will be screened with a medical history and physical examination, as well as blood tests to check general health, cholesterol levels, liver function, and the C-reactive protein (which responds to inflammation).
* Participants will not be permitted to take most prescription and over-the-counter medications that affect the immune system, including antihistamines and certain pain relievers. For 1 week before the study, participants will have a wash-out period without any of these medications.
* Participants will take rosuvastatin daily for 4 weeks, always in the evening (to ensure consistent blood sample results).
* Participants will provide blood samples at the following time points: (1) immediately before the start of the rosuvastatin treatment, (2) after 2 weeks of treatment, (3) after 4 weeks of treatment, and (4) 2 weeks after the end of treatment.

DETAILED DESCRIPTION:
Statins are drugs that inhibit cholesterol synthesis and are used extensively for primary and secondary prevention of heart disease. Their benefit to patients with heart diseases appears to exceed that predicted from cholesterol lowering alone. A recent study has found benefits of statin therapy in patients with normal cholesterol and high C-reactive protein, a marker of inflammation, suggesting that statins exert an anti inflammatory effect in addition to the well known cholesterol lowering activity. Studies in mice have revealed mixed observations regarding the role of statins in inflammation. Therefore the Center for Human Immunology, Autoimmunity and Inflammation is conducting this trial to study the effects of statins on the immune system and the inflammatory response in healthy volunteers with normal cholesterol levels, and normal or elevated C-reactive protein levels.

The primary objective is to characterize the immune system before and during statin therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Healthy volunteer (health status confirmed by brief History and Physical Exam and routine blood work as determined by the screening protocol)
* Age greater than or equal to18 years of age
* LDL < 160 mg/dL
* Ten subjects must have hsCRP < 2mg/L, and ten subjects must have hsCRP greater than or equal to 2 mg/L
* Subjects with psoriasis that are otherwise healthy, who have not received any systemic imunosuppression in the past 6 months
* Subjects with fasting glucose < 125 mg/dL

EXCLUSION CRITERIA:

* Female subjects may not be pregnant or lactating due to minor side effects of use of statins in a non-benefit study.
* Abnormal LFT s, i.e. AST > 34 U/L; ALT > 41 U/L; T. Bilirubin >1.0 mg/dL; Alkaline Phosphatasse > 116 U/L.
* Other contraindication to statins (i.e. inadequately treated hypothyroidism, renal impairment, liver disease, elevated transaminases, diabetes mellitus or hypersensitivity to a statin)
* Subjects unable to comprehend the investigational nature of the procedure or unable or unwilling to sign the consent.
* Statin usage within the last six months prior to enrollment.
* Diabetes mellitus
* Subjects not willing to participate in the gene expression analysis and whole genome expression and polymorphisms studies portion of this protocol.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-07-01; Study Completion 2018-10-04

PRIMARY OUTCOMES:
To elucidate the effects of a four week course of statins on the immune system in healthy volunteers with normal cholesterol with or without elevated C- reactive protein.
  An understanding of the mechanism by which statins effect the immune system may help us better define the patient population that might benefit from such therapy and potentially develop drugs that act more selectively and potently on the relevant immunologic pathway(s). We will also address the potential antithrombotic activity of statins.This study has been slow to recruit healthy subjects with elevated CRP, often because subjects with elevated CRP had mild abnormalities on a detailed history and physical exam, such as impaired fasting glucose. In addition, preliminary analysis of the cohort of normal CRP suggests a significant reduction in serum IL-17 during statin therapy. Psoriasis is an inflammatory disease that affects the skin and the joints, is assumed to be IL-17 driven17, and subjects are usually free of systemic imunosuppression.

SECONDARY OUTCOMES:
To describe the effects of statins on platelet activity and coagulation during thrombus formation.

CONTACTS AND LOCATIONS:
Overall Officials: Angelique Biancotto, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Karmaus PW, Shi M, Perl S, Biancotto A, Candia J, Cheung F, Kotliarov Y, Young N, Fessler MB; CHI Consortium. Effects of rosuvastatin on the immune system in healthy volunteers with normal serum cholesterol. JCI Insight. 2019 Nov 1;4(21):e131530. doi: 10.1172/jci.insight.131530. PMID 31573980